CLINICAL TRIAL: NCT00843180
Title: Massage for Children Undergoing Bone Marrow Transplantation
Brief Title: Massage for Pediatric Oncology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H41337-33343
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Results first posted 2012-05-02 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Bone Marrow Transplantation; Distress
Keywords: Bone Marrow Transplant; Massage; Pediatric Oncology; children undergoing bone marrow transplantation
MeSH Terms: interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- massage (Experimental)
  Interventions: Other: massage
- control (No Intervention): usual care only as control arm

INTERVENTIONS:
Other: massage — one to three massages per week by massage practitioner additional massages by resident parent who is being taught to massage her/his child
  Arms: massage

SUMMARY:
Undergoing bone marrow transplantation (BMT) is associated with a high level of distress for patients and caregivers. Clinical research studies have reported benefits from massage for a) oncology patients, b) children, c) adults and children undergoing bone marrow transplants. A multi-center study of an intervention using a combination of massage therapy and a laugh cart to reduce distress in pediatric oncology patients undergoing BMT (PI: Phipps) is completed with results not yet published. There is still a need for independent studies to isolate the effect of massage for clinical outcomes (such as improved nausea and pain control) in children. Furthermore, this study will test the acceptability of an augmented massage intervention. In addition to provider-child massage, the augmented massage intervention includes training of the resident parent to provide additional parent-child massage, to relieve symptoms as needed. The goal of this augmented intervention is the improvement of symptom management in patients and decreased stress and feelings of helplessness in parents.

We propose a randomized pilot study at the UCSF pediatric bone marrow transplant center to assess the feasibility of a higher-quality study of the effects of massage in this population.

Aim 1: Determine the acceptability of a massage intervention for patients and parents on a pediatric bone marrow transplant unit.

Aim 2: Explore the logistics of implementing the augmented massage intervention at the bedside offered to consecutive patients over one year's time.

Aim 3: Collect preliminary data for patients and parents including patient clinical outcomes, quality of life, and satisfaction, and parental stress and mood to allow sample size calculations for further studies.

DETAILED DESCRIPTION:
This study is a pilot randomized controlled feasibility trial of an augmented massage intervention, compared to a usual-care control group, in which intervention group participants will receive up to 3 massage sessions per week, during the 4-6 hospitalization at UCSF for Bone Marrow Transplant (BMT).

Participants will be approximately 24 children recruited from consecutive sample of pediatric cancer and non-cancer patients undergoing BMT age 5 to 18 admitted to UCSF children's hospital during one calendar year.

Intervention: Massage sessions will be gentle Swedish style combine with acupressure and will range from 20-45 minutes, provided by credentialed and trained massage therapists; augmentation will involve massage training for the resident parent, who rooms with the patient, to administer massage to his/her child during the course of the hospital stay. The control group will receive standard-care.

We will collect feasibility data and do exploratory comparison of clinical outcomes between groups.

Knowledge to be gained: We will have preliminary data for a larger trial that will determine whether an augmented massage intervention can support symptom management in the pediatric BMT unit.

B. Hypothesis(es): Briefly explain the hypothesis(es) to be tested. If the study is not designed to test a hypothesis, simply state "None." Hypothesis 1a: >60% of Patients are willing to be randomized to the massage study.

Hypothesis 1b: 80% of patients randomized to massage will accept the massage intervention when offered.

Hypothesis 1c: The majority of parents (>60%) are willing to learn massage techniques for use on their children.

Hypothesis 2a: Professional massage providers will be able to deliver massage, negotiating schedule, space, time, and other patient-related medical activities and will be able to schedule >50% of planned massages.

Hypothesis 2b: Massage providers will be able to assess the acceptable time period for massage (between 10 minutes and 45 minutes).

Hypothesis 2c: Parents will carry out the massage on their children, will do at least 5 massages over the study period and are willing to provide a self-report of estimated time engaged in massage.

Hypothesis 3a: 80% of patients will answer survey questions about their experience in general and the massage intervention.

Hypothesis 3b: The RA will be able to collect clinical data from chart review and electronically stored lab data .

Hypothesis 3c: 80% of parents will answer survey questions about their experience in learning and delivering massage, stress, mood, PTSD symptoms and self-efficacy around patient management.

ELIGIBILITY:
Inclusion Criteria:

* Being 5 to 18 years old
* Admitted for BMT.

Rationale: This is a pediatric study for children up to age 18 admitted to the BMT unit. Questionnaires are not designed for children under age 5.

Exclusion Criteria:

* Parent or child unable to answer questionnaire due to language limitations.

Rationale: The pilot character of the study with its limited budget does not include instruments in foreign languages, such as Chinese or Spanish. This could be a project for further studies.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2008-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolf E Mehling, MD, Study Director — University of California, San Francisco
Locations (1):
- Childrens' Hospital UCSF, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: November 2008-November 2009, 12 months UCSF Children's Hospital, Bone Marrow Transplant Unit
Pre-assignment Details: consecutive enrollment of all eligible admitted children. 2 teenage boys declined participation
Groups:
- Massage: massage and acupressure up to 3x/week for entire hospital stay
- Control: usual care only as control arm hospital care during bone marrow transplant
Period: Overall Study
Arm/Group | Massage | Control
Started | 16 | 7
Completed | 16 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Massage | Control | Total
Number analyzed (Participants) | 16 | 7 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 7 | 23
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 10.9 (3.7) | 13.7 (4.3) | 11.7 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 9 | 4 | 13
Region of Enrollment [Number; unit: participants]
  United States | 16 | 7 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Days With Pain Scores >3 Measured on Numeric Rating Scale (Range 0-10; 0 for no Pain; 10 for Worst Pain Imaginable)
Description: days of pain >3 by nurses notes based on pain scores on numeric rating scale (up to 28 days)
Time Frame: 7 days pre to 21 days post transplant = 28 days
Population: ITT no imputations
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Massage | Control
Number analyzed (Participants) | 16 | 7
days | 7.7 (4.9) [5.2 to 10.2] | 8.3 (5.5) [2.8 to 13.7]
Statistical Analysis 1: Comparison: Massage vs Control; comparison between groups by t-test; Test type: Superiority or Other; p = 0.80, t-test, 2 sided — unadjusted; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-5.4 to 4.2], Standard Deviation 0 — this was a feasibility pilot study CI is descriptor of dispersion

2. Secondary Outcome: Number of Vomiting Episodes
Description: number of vomiting episodes as reported by nurses per occurence (no upper limit)
Time Frame: day -7 to +21 around transplant date
Population: ITT
Measure: Mean (95% Confidence Interval); unit: number of episodes
Arm/Group | Massage | Control
Number analyzed (Participants) | 16 | 7
number of episodes | 4.6 [2.0 to 7.3] | 7.0 [3.0 to 11.0]
Statistical Analysis 1: Comparison: Massage vs Control; Test type: Superiority or Other; p = 0.29, t-test, 2 sided — unadjusted; Mean Difference (Final Values) = -2.38, 95% CI 2-sided [-6.9 to 2.1], Standard Deviation 0 — CI serves as dispersion measure

3. Secondary Outcome: Days of Hospital Stay
Description: days of hospital stay after bone marrow transplant (up to 100 days; participant observation was censored after 100 days)
Time Frame: days of hospital stay after bone marrow transplant
Population: ITT
Measure: Mean (95% Confidence Interval); unit: number of days
Arm/Group | Massage | Control
Number analyzed (Participants) | 16 | 7
number of days | 39.1 [24.8 to 53.3] | 35.3 [2.1 to 68.4]
Statistical Analysis 1: Comparison: Massage vs Control; Test type: Superiority or Other; p = 0.78, t-test, 2 sided; Median Difference (Final Values) = -3.8, 95% CI 2-sided [-31.9 to 24.3], Standard Deviation 0 — 95% CI is dispersion parameter

4. Secondary Outcome: Days to Recovery Neutrophil Count
Description: number of days to recovery neutrophil count >500 cells per microliter for 2 consecutive days (range, up to 100 days, censored at 100 days)
Time Frame: hospital stay
Measure: Mean (95% Confidence Interval); unit: number of days
Arm/Group | Massage | Control
Number analyzed (Participants) | 16 | 7
number of days | 16.8 (14.3) [14.3 to 19.4] | 18.7 [7.3 to 30.0]
Statistical Analysis 1: Comparison: Massage vs Control; Test type: Superiority or Other; p = 0.70, t-test, 2 sided; unadjusted; Mean Difference (Final Values) = 5.8, 95% CI 2-sided [-9.5 to 13.2], Standard Deviation 0 — 95%CI is dispersion measure

ADVERSE EVENTS:
Time Frame: any adverse events were documented during entire hospital stay, censored at 100 days.
Description: Medical records were checked weekly, nurse managers were contacted regularly, attending physicians were ready to inform the research team for any eventual adverse events.
Arm/Group | Massage | Control
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/7
Other Adverse Events (participants affected / at risk) | 0/16 | 0/7

LIMITATIONS AND CAVEATS:
1. small sample size
2. limited number of time points for self-report assessments.
3. the dose of the massage intervention averaged 1.8 massages per week, while the target dose was 3 per week.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No